CLINICAL TRIAL: NCT04328948
Title: A Randomized Controlled Phase III Trial of Comparing Local Field With Additional Prophylactic Irradiation in Chemoradiotherapy for Clinical-T1bN0M0 Esophageal Cancer
Brief Title: A Randomized Controlled Trial Evaluating of Prophylactic Irradiation in CRT for cT1bN0M0 ESCC
Acronym: ARMADILLO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Responsible Party: Principal Investigator, Ken Kato, National Cancer Center Hospital, National Cancer Center, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1904
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; chemoradiotherapy; Radiation Field
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemoradiation therapy with elective nodal irradiation (Experimental): Chemoradiotherapy consists of 5-FU (1,000 mg / m2, day1-4, day29-32), CDDP (75 mg /m2, day1, 29) and radiotherapy (50.4 Gy/28Fr)
  Interventions: Radiation: Chemoradiotherapy
- Chemoradiation therapy with involved field irradiation (Active Comparator): Chemoradiotherapy consists of 5-FU (700 mg /m2, day1-4, day29-32), CDDP (70 mg /m2, day1,29) and radiotherapy (60 Gy/30Fr)
  Interventions: Radiation: Chemoradiotherapy

INTERVENTIONS:
Radiation: Chemoradiotherapy — Chemoradiotherapy

SUMMARY:
This study is conducted to investigate whether modified chemoradiotherapy with elective nodal irradiation reduces the locoregional recurrence that cannot be completely resected by salvage endoscopic resection and preserve esophagus without compromising overall survival.

ELIGIBILITY:
Inclusion criteria:

1. Histologically proven squamous cell carcinoma, adenosquamous carcinoma, or basaloid cell carcinoma.
2. All lesions located in the thoracic esophagus. Secondary lesions with an absolute indication for endoscopic resection (EMR/ESD) may not be confined to the thoracic esophagus.
3. Clinical N0M0 with cervical to abdominal contrast-enhanced CT.
4. The deepest lesion is diagnosed as cT1b (SM1 / SM2 / SM3) with upper gastrointestinal endoscopy. If it is difficult to differentiate cT1a-MM and cT1b-SM1 clinically, the wall depth is diagnosed as cT1b-SM1.
5. Aged 20 years and older.
6. ECOG Performance status 0 or 1.
7. No previous therapy against esophageal cancer except for complete resection by EMR/ESD with either pT1a-LPM (pM2) / pT1a-MM (M3) disease or pT1a-MM (M3) disease without vascular infiltration.
8. No history of radiotherapy for the neck, chest, and upper abdomen for any cancers. No chemotherapy or hormone therapy with less than 3 years of disease-free interval for any cancers.
9. Major organ function is preserved. 1) WBC<=12,000/mm3 2) ANC>=1,500/mm3 3) Hb>=10.0 g /dL 4) PLT>=10,000/mm3 5) T-bil<=1.5 mg /dL 6) AST<=100 IU/L 7) ALT<=100 IU/L 8) SpO2>=95% 9) Ccr>=60 mL/min
10. Patients do not have a preference to receive a surgical resection as an initial therapy after receiving explanations.
11. Written informed consent is obtained.

Exclusion criteria:

1. Simultaneous or metachronous (within 5 years) double cancers, except for intramucosal tumor curable with local therapy.
2. Active infection requiring systemic therapy.
3. Fever over 38 degrees Celsius
4. Female during pregnancy, within 28 days of post parturition, or during lactation. Male who wants a partner's pregnancy.
5. Psychological disorder, which is difficult to participate in this clinical study.
6. Receiving continuous systemic corticosteroid or immunosuppressant treatment.
7. Positive for HBs antigen or HIV antigen.
8. Diabetes mellitus, which is uncontrollable with continuous use of insulin or hypoglycemic agents.
9. Uncontrolled arterial hypertension.
10. History of unstable angina pectoris within three weeks or myocardial infarction within six months before registration.
11. Uncontrolled valvular disease, dilated cardiomyopathy, and hypertrophic cardiomyopathy.
12. Severe emphysema, interstitial pneumonia or pulmonary fibrosis based on chest CT.
13. With a history of cerebrovascular disorder within 6 months.
14. Drug allergy for iodic drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Major progression-free survival | The primary analysis will be held 5-years after the last patient was enrolled.
  If the remnant lesion in the esophagus or a recurrent lesion after complete response (CR) can be curatively removed by salvage EMR/ESD, it is not an event, and other progressions and deaths are events.

SECONDARY OUTCOMES:
Overall survival | The primary analysis will be held 5-years after the last patient was enrolled.
  From date of randomization to date of death, approximately 5 years.
Progression-free survival | The primary analysis will be held 5-years after the last patient was enrolled.
  From date of randomization to date of progression or death, whichever occurs first, approximately 5 years.
Complete response rate | The primary analysis will be held 5-years after the last patient was enrolled.
  CR was defined as disappeared primary tumors without the presence of ulceration or malignant cells in biopsy specimens under endoscopy.
Esophagectomy-free survival | The primary analysis will be held 5-years after the last patient was enrolled.
  From date of randomization to date of esophagectomy or death, whichever occurs first, approximately 5 years.
Adverse events | The primary analysis will be held 5-years after the last patient was enrolled.
  Number of participants with treatment-related adverse events during CRT as assessed by CTCAE v4.0
Long term toxicity | The primary analysis will be held 5-years after the last patient was enrolled.
  Number of participants with treatment-related adverse events after termination of CRT as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kato, MD/PhD, Study Chair — National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided